CLINICAL TRIAL: NCT03924908
Title: Impact of Virtual Reality Hypnosis on Pain and Anxiety During Dressings Change in Burn Patients Treated as Outpatients
Brief Title: Impact of Virtual Reality Hypnosis on Pain and Anxiety During Dressings Change in Burn Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough human resources
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, Head of Clinic, principal investigator, University of Liege
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BurnVR-H
Record Dates: First submitted 2019-04-11; First posted 2019-04-23 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Burns; Pain, Acute; Anxiety
MeSH Terms: conditions — Burns; Acute Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRH (Experimental): Virtual reality hypnosis
  Interventions: Behavioral: VRH
- VR (Active Comparator): Virtual reality
  Interventions: Behavioral: VR

INTERVENTIONS:
Behavioral: VRH — Patients will see a 3D film combined with a hypnotic voice during the entire procedure of dressing change
  Arms: VRH
Behavioral: VR — Patients will see a 3D film without any hypnotic voice during the entire procedure of dressing change
  Arms: VR

SUMMARY:
Different non-pharmacological techniques, including hypnosis and virtual reality are currently used as complementary tools in the treatment of pain related to burn injury. A new technique called 'virtual reality hypnosis' (VRH) (Patterson et al., 2004), which encompasses a combination of both tools, is regularly used although its actual function remains unknown to this date. With the goal to improve our understanding of VRH combination effects, it is necessary to elaborate randomized and controlled research studies in order to understand their actual function in individual's perception. 100 patients who are treated as outpatients for burn care will be randomly assigned to virtual reality or VRH. Patients will receive one session of one of these techniques during burn dressing change.Physiological parameters will be recorded during dressing change. Participants will fill in a questionnaire evaluating their tendency to be absorbed and dissociated, and another evaluating their level of perceived immersion. Their level of anxiety, pain, fatigue and relaxation will be evaluated before and after the session. A short interview will also be conducted to give participants the opportunity to openly describe their experience.

ELIGIBILITY:
Inclusion Criteria:

* Burn patient treated as outpatient
* Burn surface area > or = 5% of the total body surface area
* mainly 2nd degree burn

Exclusion Criteria:

* Psychiatric antecedents
* Claustrophobia
* Heavy hearing
* Visual impairment
* Face burn
* Conjunctivitis
* Consent not obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain perception: Visual Analogical Scale (VAS) | 5 minutes before dressing change ("time 0") and 5 minutes after dressing change ("time 1")
  Visual Analogical Scale (VAS) from 0 to 10. This is a subjective linear scale. No pain = 0, maximum pain = 10.
Change in anxiety: Visual Analogical Scale (VAS) | 5 minutes before dressing change ("time 0") and 5 minutes after dressing change ("time 1")
  Visual Analogical Scale (VAS) from 0 to 10. This is a subjective linear scale. No anxiety = 0, maximum anxiety = 10.
Change in fatigue | 5 minutes before dressing change ("time 0") and 5 minutes after dressing change ("time 1")
  Visual Analogical Scale (VAS) from 0 to 10. This is a subjective linear scale. No fatigue = 0, maximum fatigue = 10.
Change in relaxation level | 5 minutes before dressing change ("time 0") and 5 minutes after dressing change ("time 1")
  Visual Analogical Scale (VAS) from 0 to 10. This is a subjective linear scale. No relaxation = 0, maximum relaxation = 10.

SECONDARY OUTCOMES:
Level of absorption at the moment | 5 minutes after dressing change ("time 1")
  Absorption will be measured as the two components of hypnosis. We will measure absorption and dissociation using the Visual Analogical Scales (VAS). VAS is from 0 to 10. 0 is not absorbed and 10 is really absorbed. When responding to a VAS item, participants will be asked to specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Level of dissociation at the moment | 5 minutes after dressing change ("time 1")
  Dissociation will be measured as the two components of hypnosis. We will measure absorption and dissociation using the Visual Analogical Scales (VAS). When responding to a VAS item, participants will be asked to specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Time perception | 5 minutes after dressing change ("time 1")
  We will ask to the patient his perception of time during the session.
Change in heart rate | 5 minutes before dressing change ("time 0") and 5 minutes after dressing change ("time 1")
  Physiological parameter measured using pulse oximeter

OTHER OUTCOMES:
Participant's tendency to be absorbed and dissociated | At inclusion (Day -2)
  Tellegen Absorption Scale (TAS). Participants answer "true" or 'false" at each items (34). The subject's score is simply the number of items marked "true".
Participant's opinion about the tool | 5 minutes after dressing change ("time 1")
  Satisfaction questionnaire created by our lab to understand if patients have a good adherence about the tool or not. Some items should be marked as "yes" or "not" and some items are marked from 1 ("not at all") to 7 ("enormously")

IPD SHARING:
Plan to Share IPD: No